CLINICAL TRIAL: NCT04070651
Title: Sleep Disturbance and Its Association With Fatigue, Depressive Symptoms, and Clinical Response to Immune Checkpoint Inhibitors (ICI) in Lung Cancer Patients
Brief Title: Sleep and Immune Checkpoint Inhibitors
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Louise Strøm, PhD-fellow, University of Aarhus
Other Study IDs: Sleep.ICI
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer
Keywords: Sleep; Fatigue; Depressive symptoms; Immune Checkpoint Inhibitors; Lung Cancer; Clinical response
MeSH Terms: conditions — Lung Neoplasms; Fatigue; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sleep disturbances are prevalent in cancer patients and linked to levels of fatigue and depressive symptoms with a major impact on quality of life. A growing body of evidence links sleep disturbances with various health outcomes, including increased risk of depression, cancer, and overall mortality. Inflammation is suggested to be an underlying mechanism both driving and maintaining the symptom cluster of sleep disturbance, fatigue and depressive symptoms, as well as being bi-directionally linked to sleep. The main purpose of the present study is to investigate the prevalence of sleep disturbance and its association with psychological and physical symptoms as well as the clinical response to ICI in non-small-cell lung cancer patients (NSCLC), with a secondary aim of exploring the role of inflammation.

DETAILED DESCRIPTION:
A total of 240 cancer patients diagnosed with advanced NSCLC, referred to treatment with ICI will be enrolled in this prospective observational study. Patients will be assessed prior to initiation of treatment (baseline) and every third subsequent week, corresponding to each treatment cycle over a period of 18 weeks. Assessments will include questionnaires, sleep diaries, actigraphy, and blood and saliva samples to examine sleep, fatigue, psychological and physical symptoms, the sleep-wake-cycle, inflammation, and cortisol. Additionally, the patients will be asked to complete a reduced questionnaire every week within the 18 weeks period, to address weekly fluctuations in sleep quality, fatigue, and mood. Treatment response is assessed after 9 and 18 weeks.

Aims:

1. To explore possible associations between sleep and the clinical response to treatment with ICI.
2. To investigate the prevalence of sleep disturbance in patients with NSCLC during treatment with ICI.
3. To prospectively assess changes in sleep parameters over the course of treatment.
4. To examine associations between sleep parameters and fatigue, depression, anxiety, and inflammation.
5. To explore possible associations between sleep, fatigue, depression, inflammatory responses and the clinical response to treatment with ICIs.

Hypotheses:

Patients with high levels of sleep disturbance (insomnia severity) will experience 1) poorer clinical response to ICI, 2) more depressive symptoms, 3) higher levels of fatigue, 4) poorer overall health-related quality of life (HRQoL), 5) higher levels of inflammation.

ELIGIBILITY:
Inclusion Criteria:

- Confirmed diagnosis of advanced non-small cell lung cancer

Exclusion Criteria:

* Insufficient Danish proficiency
* Pre-existing confounding psychiatric illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women diagnosed with advanced non-small cell lung cancer, treated with immune checkpoint inhibitors, at Aarhus University Hospital, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Clinical response to treatment | Changes from baseline to 9 and 18 weeks after treatment initiation, respectively.
  Radiological evaluation of the clinical response to treatment with ICI, according to RECIST criteria.

SECONDARY OUTCOMES:
Insomnia Severity | Weekly from baseline to 18 weeks after treatment initiation, and follow-up 1, 2 and 3 years from baseline, respectively.
  Changes in insomnia severity as measured with The Insomnia Severity Index (ISI). Total score ranges from 0 to 28. Interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Sleep diary | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively.
  Changes in Standard sleep metrics (nightly sleep onset latency (SOL), wakefulness after initial sleep onset (WASO), total sleep time (TST), total time spent in bed (TIB), sleep efficiency (SE).
Fatigue | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively, and follow-up 1, 2 and 3 years from baseline, respectively.
  Changes in subjective fatigue as measured with the Multidimensional Fatigue Symptom Inventory - Short Form (MFSI-SF). Subscales (general, physical, emotional, and mental fatigue) are summed and the vigor scale subtracted to create a fatigue total score, with higher scores indicating higher levels of fatigue.
Depressive symptoms | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively, and follow-up 1, 2 and 3 years from baseline, respectively.
  Changes in depressive symptoms as measured with the Patient-Reported Outcomes Measurement Information System (PROMIS®) Depression - Short Form 8a. Total raw score ranges from 8 to 40, with higher scores indicating greater severity of depression.
Health-related quality of life | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively, and follow-up 1, 2 and 3 years from baseline, respectively.
  Changes in health-related quality of life as measured with The European Organization for Research and Treatment of Cancer, Quality of Life questionnaire for cancer patients (EORTC QLQ-C30). The standardized raw score, ranges from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Disease specific health-related quality of life | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively, and follow-up 1, 2 and 3 years from baseline, respectively.
  Changes in disease specific health-related quality of life as measured with The European Organization for Research and Treatment of Cancer, Quality of Life Lung Cancer Module (EORTC QLQ-LC29). The standardized raw score, ranges from 0 to 100; a high score for the symptom scales / single items represents a high level of symptomatology or problems.
Perceived Stress | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively, and follow-up 1, 2 and 3 years from baseline, respectively.
  Changes in perceived stress as measured with The Perceived Stress Scale (PSS). Total score ranges from 0 to 40, with higher scores indicating higher perceived stress.
Sickness behavior | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively, and follow-up 1, 2 and 3 years from baseline, respectively.
  Changes in subjective sickness behavior as measured with the Sickness Questionnaire (SicknessQ). Total score ranges from 0 to 30, with higher scores indicating more sickness behaviour.
Cortisol | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively.
  Cortisol awakening response (CAR), and the diurnal cortisol slope (DCS)
Inflammatory response 1 | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively.
  CRP
Inflammatory response 2 | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively.
  IL-6
Inflammatory response 3 | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively.
  TNF-a
Inflammatory response 4 | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively.
  Se-Cortisol
Inflammatory response 5 | Baseline, and week 3, 6, 9, 12, 15 and 18, respectively.
  White blood cell count.
Actigraphy 1 | Baseline to 18 weeks after initiation of treatment.
  Objective sleep outcome. Nightly sleep onset latency (SOL)
Actigraphy 2 | Baseline to 18 weeks after initiation of treatment.
  Objective sleep outcome: Wakefulness after initial sleep onset (WASO)
Actigraphy 3 | Baseline to 18 weeks after initiation of treatment.
  Objective sleep outcome: Total sleep time (TST)
Actigraphy 4 | Baseline to 18 weeks after initiation of treatment.
  Objective sleep outcome: Total time spent in bed (TIB)
Actigraphy 5 | Baseline to 18 weeks after initiation of treatment.
  Objective sleep outcome: Sleep efficiency (SE, i.e., the percent of the time asleep out of amount of time spent in bed)
Actigraphy 6 | Baseline to 18 weeks after initiation of treatment.
  Objective sleep outcome: Circadian activity rhythms.
Disease status | 1, 2 and 3 years from treatment initiation (baseline).
  Changes in disease status after treatment initiation with ICI. Changes are evaluated according to RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zachariae, Prof., DMSc, Study Director — Aarhus University and Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided